CLINICAL TRIAL: NCT05703958
Title: An Open Label, Multi-Center, Retrospective and Prospective Evaluation of Equinoxe Proximal Humerus Fracture Plates Clinical and Radiographic Outcomes
Brief Title: Exactech Proximal Humerus Fracture Plate System Post Market Clinical Follow-up
Status: Recruiting | Type: Observational
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Other Study IDs: CR21-001
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Proximal Humeral Fracture; Fracture Dislocation; Non-Union Fracture
MeSH Terms: conditions — Shoulder Fractures; Fracture Dislocation; Fractures, Ununited

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to collect and evaluate long-term clinical outcomes data in order to better understand the safety and performance of the Equinoxe Proximal Humerus Fracture Plates over time. This study will follow subjects for a period of up to 10 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated to receive Equinoxe Proximal Humerus Fracture Plate or has previously underwent primary surgery with Equioxe Proximal Humerus Fracture Plate
* Patient is willing to participate by complying with pre- and postoperative visit requirements
* Patient is willing to agree to be followed for up to 10 years following their index surgery
* Patient is willing and able to review and sign a study informed consent form

Exclusion Criteria:

* Osteomyelitis of the proximal humerus or scapula
* Inadequate or malformed bone that precludes adequate support or fixation of the prosthesis
* Patient's age, weight, or activity level would cause the surgeon to expect early failure of the system
* The patient is unwilling or unable to comply with the post-operative care instructions
* Alcohol, drug, or other subtance abuse
* Any disease state that could adversaly affect the function or longevity of the implant
* Patient is pregnant
* Patient is a prisoner
* Patient has a physical or mental condition that would invalidate the results

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ORIF surgery who meet eligibility criteria - Patients who consent to participate to return for follow-up visits out to 10 years or longer
Sampling Method: Non-Probability Sample
Enrollment: 151 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2034-09-30 (Estimated)

PRIMARY OUTCOMES:
Smart Score | Through study completion, an average of 1 per year
  Shoulder Arthroplasty Smart (SAS) score - 6 questions based on 3 objective active range of motion and 3 subjective measures of pain and function. Score range of 0 to 100 where 100 indicates the best score
Sane Score | Through study completion, an average of 1 per year
  Single Assessment Numeric Evaluation (SANE) - Patient shoulder self-evaluation as a percentage of normal, 100% corresponds being normal
ASES | Through study completion, an average of 1 per year
  American Shoulder and Elbow Surgeons Score (ASES) - 100 points scale about shoulder pain and performance evaluation in activities of daily living where 100 indicates the best shoulder condition
Quick DASH | Through study completion, an average of 1 per year
  Shorten version of Disability of the Arm, Shoulder, and Hand (DASH) - 11 items to measure ability of a patient to perform certain upper extremity where 0 corresponds to no difficulty and 100 corresponds to unable

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Ganta, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Grossman School of Medicine, New York, New York, United States